CLINICAL TRIAL: NCT01259375
Title: A Phase II Study of Amrubicin Chemotherapy as First Line Treatment in Patients With Metastatic or Unresectable Soft Tissue Sarcoma
Brief Title: Amrubicin Chemotherapy as First Line in Metastatic or Unresectable Soft Tissue Sarcoma
Acronym: ARSARC-PI-0010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI45197
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All participants who received Amrubicin.
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Amrubicin — Synthetic 9-aminoanthracycline Patients will receive 40mg/m2/day intravenously

SUMMARY:
Primary Objectives

1. To evaluate the Response Rate (RR) for amrubicin in patients with metastatic or advanced sarcoma as first line therapy.
2. To evaluate Progression Free Survival (PFS).

Secondary Objectives

1. To assess the safety and tolerability of amrubicin in this patient population.
2. To evaluate whether certain histologic subtypes of sarcoma demonstrate a differential response to amrubicin.
3. To investigate quality of response with radiographic evaluation using both Response Evaluation Criteria In Solid Tumors (RECIST) and Choi criteria.
4. To evaluate overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older)
* Pathological diagnosis of soft tissue sarcoma. Pathology materials must be submitted and reviewed.
* Patients must have unresectable locally advanced or metastatic progressive disease prior to enrollment. Disease extent must be determined by scans (CT or PET CT) within 6 weeks of enrollment.
* No prior chemotherapy for soft tissue sarcoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function including the following:
* Adequate bone marrow reserve: absolute neutrophil count (segmented and bands) (ANC) 1.5 x 109/L, platelet count 100 x 109/L, and hemoglobin 90 g/L,
* Hepatic: bilirubin 1.5 x the upper limit of normal (ULN), ALT and AST 3.0 x ULN,
* Renal: serum creatinine 1.5 x ULN or calculated creatinine clearance greater than 60 mL/min,
* Cardiac: Left ventricular ejection fraction (LVEF) 50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA);
* All labs must be done within 2 weeks prior to enrollment.
* Negative serum pregnancy test at the time of enrollment for females of childbearing potential;
* For males and females of child-producing potential, use of effective contraceptive methods during the study;
* Ability to understand the requirements of the study and provide written informed consent.

Exclusion Criteria:

* Pregnant or nursing females
* Chest radiotherapy with curative intent to the primary disease complex less than or equal to 28 days prior to first dose; cranial radiotherapy less than or equal to 21 days prior to first dose; radiotherapy to all other areas less than or equal to 7 days prior to first dose
* Concurrent severe or uncontrolled medical disease (eg, active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure, active viral hepatitis or chronic liver disease) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study
* Symptomatic central nervous system metastases. Patients with asymptomatic brain metastases are allowed. The patient must be stable for 2 weeks after radiotherapy; if the patient is on corticosteroids, the dose of corticosteroids must have been stable for 2 weeks prior to first dose of study treatment, or be in the process of being tapered
* Suspected, diffuse idiopathic interstitial lung disease or pulmonary fibrosis.
* Patients with known history of seropositive human immunodeficiency virus (HIV) or patients who are receiving immunosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications. HIV testing is not required for inclusion in the trial.
* Known hypersensitivity to any of the components of the i.v. formulation of amrubicin.
* Psychiatric disorder or any other personal circumstances that prevent compliance with the study protocol.
* Inability or unwillingness to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Santa Monica, Santa Monica, California
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All participants enrolled.
  Amrubicin: Synthetic 9-aminoanthracycline Patients will receive 40mg/m2/day intravenously
Period: Overall Study
Arm/Group | All Patients
Started | 24
Completed | 23
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- All Groups: All patients that received treatment.
Arm/Group | All Groups
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 52 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for Amrubicin in Patients With Metastatic or Advanced Sarcoma as First Line Therapy.
Description: Per response evaluation criteria in solid tumors criteria (RECIST 1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 48 months
Population: One patient discontinued study treatment after the first cycle due to side effects and was not evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of pt with a partial response
Arm/Group | All Patients
Number analyzed (Participants) | 23
percentage of pt with a partial response | 13 [2.8 to 33.6]

2. Primary Outcome: Progression Free Survival
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.1) for target lesions and assessed by CT; time elapsed between treatment initiation and tumor progression or death. In target lesions, progression is defined per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1) as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. In non-target lesions, progression is defined via RECIST v 1.1 as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: six months
Measure: Number (95% Confidence Interval); unit: percentage of pt with 6 mnth PFS
Arm/Group | All Patients
Number analyzed (Participants) | 23
percentage of pt with 6 mnth PFS | 42.7 [24.0 to 76.3]

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Time Frame: 4 months
Population: One patient discontinued study treatment after the first cycle due to side effects and was not evaluable for response, but was evaluable for safety and toxicity.
Measure: Number; unit: participants who experienced an SAE
Arm/Group | All Patients
Number analyzed (Participants) | 24
participants who experienced an SAE | 7

4. Secondary Outcome: Overall Survival
Description: This variable reviews the percentage of Overall Survival at 24 months and presents the percentage of participants who survived at 2 years.
Time Frame: two years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 23
percentage of participants | 52.8 [35.9 to 77.6]

5. Secondary Outcome: Quality of Response With Radiographic Evaluation Using Both Response Evaluation Criteria In Solid Tumors (RECIST) and Choi Criteria.
Description: Per response evaluation criteria in solid tumors criteria (RECIST 1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Exploratory CT evaluations according to Choi response criteria will be also performed and correlated with RECIST response.
Time Frame: 48 months
Population: This exploratory objective was not assessed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Differential Response to Amurbicin Among Certain Histologic Subtypes of Sarcoma.
Description: as for outcome 1
Time Frame: 48 months
Measure: Number; unit: participants
Groups:
- All Groups: All patients who had a partial or greater response
Arm/Group | All Groups
Number analyzed (Participants) | 3
participants
  liposarcoma | 1
  myxoid liposarcoma with TLS-CHOP translocation | 1
  leiomyoscarcoma | 1

ADVERSE EVENTS:
Time Frame: Through study treatment, an average of 4 months.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=24)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
febrile neutropenia (Blood and lymphatic system disorders) | 4
back pain (Musculoskeletal and connective tissue disorders) | 1
e. coli positive (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=24)
abdominal discomfort (Gastrointestinal disorders) | 2
abdominal pain (Gastrointestinal disorders) | 2
Agitation (Psychiatric disorders) | 2
alopecia (Skin and subcutaneous tissue disorders) | 21
anemia (Blood and lymphatic system disorders) | 6
anorexia (Metabolism and nutrition disorders) | 8
back pain (Musculoskeletal and connective tissue disorders) | 3
blurred vision (Eye disorders) | 2
body aches (Musculoskeletal and connective tissue disorders) | 2
chills (General disorders) | 2
congestion (Respiratory, thoracic and mediastinal disorders) | 3
constipation (Gastrointestinal disorders) | 4
cough (Respiratory, thoracic and mediastinal disorders) | 11
despression (Psychiatric disorders) | 2
diarrhea (Gastrointestinal disorders) | 4
dry eyes (Eye disorders) | 2
dry skin (Skin and subcutaneous tissue disorders) | 2
dysgeusia (Gastrointestinal disorders) | 5
dyspenia (Respiratory, thoracic and mediastinal disorders) | 5
edema (General disorders) | 4
fatigue (General disorders) | 18
fever (General disorders) | 5
headaches (Nervous system disorders) | 6
hiccups (Respiratory, thoracic and mediastinal disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 2
hypertension (Cardiac disorders) | 2
hypoalbuminemia (Metabolism and nutrition disorders) | 2
insomnia (Psychiatric disorders) | 5
neutropenia (Blood and lymphatic system disorders) | 5
oral thrush (Gastrointestinal disorders) | 2
thrombocytopenia (Blood and lymphatic system disorders) | 3
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 3
reflux (Gastrointestinal disorders) | 7
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4
Sinus bradycardia (Cardiac disorders) | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4
vomiting (Gastrointestinal disorders) | 5
weight loss (Investigations) | 2
white blood cell decreased (Investigations) | 5
decreased joint function (Musculoskeletal and connective tissue disorders) | 2
malaise (General disorders) | 2
mucositis (Respiratory, thoracic and mediastinal disorders) | 5
myalgia (Musculoskeletal and connective tissue disorders) | 2
nausea (Gastrointestinal disorders) | 17
mouth sores (Gastrointestinal disorders) | 2
hip pain (Musculoskeletal and connective tissue disorders) | 2
lower extremity pain (Musculoskeletal and connective tissue disorders) | 3
tachycardia (Cardiac disorders) | 3
gait disturbance (General disorders) | 2
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No